CLINICAL TRIAL: NCT04841070
Title: NEURodevelopmental Outcome in Children Between One and Five Years After Persistent Pulmonary Hypertension Of the Newborn
Brief Title: NEURodevelopmental Outcome After Persistent Pulmonary Hypertension Of the Newborn
Acronym: NEUROPHON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0186
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Glycation End Products, Advanced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persistent pulmonary hypertension of the newborn. (Experimental): Children aged 1 to 5 years who have been hospitalized in pediatric resuscitation service for the treatment of persistent pulmonary hypertension of the newborn.
  Interventions: Other: Ages & Stages Questionnaires®, Third Edition (ASQ3)

INTERVENTIONS:
Other: Ages & Stages Questionnaires®, Third Edition (ASQ3) — Investigators will propose to parents of children hospitalized for the treatment of persistent pulmonary hypertension of the newborn a hetero-evaluation via the validated ASQ questionnaire to analyze neuro-psychomotor development.

SUMMARY:
Neonatal pulmonary hypertension is a rare but serious condition resulting from a lack of adaptation to extra-uterine life in some newborns. In the short term, the risk of death requires rapid and appropriate management of this transient pathology.

In the long term, these newborns present a greater brain vulnerability, a consequence of the pathology itself with cerebral hypoxia but also invasive and aggressive therapies. Although current scientific evidence indicates a correlation with the existence of neurological developmental disorders, the understanding of the long-term neurological outcome of these babies remains poorly documented. Better knowledge of remote neuro-psychomotor development of the critical period

ELIGIBILITY:
Inclusion Criteria:

* All parenting authority holders of children aged 1 to 5 years, born after 34 weeks of amenorrhea and having been cared for neonatal PAH in paediatric resuscitation

Exclusion Criteria:

* Holders of parental authority who cannot answer the questionnaire because they do not speak French.
* Opposition of one of the two holders of parental authority
* Minor parental authority holders
* Holders of parental authority under safeguarding of justice, guardianship or guardianship
* Newborns with neonatal PAH with an associated diagnosis of diaphragmatic hernia or cyanogenic congenital heart disease
* Newborns with neonatal PAH not treated with nitrogen monoxide

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Describe the association between the occurrence of neuro-psychomotor developmental disorders and initial management in resuscitation. | Between one and 5 years after hospitalization in resuscitation.
  Parents will complete ASQ3. The investigators will consider neuro-psychomotor developmental disorders in children with pathological ASQ questionnaire on at least 2 items.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BREINIG, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France